CLINICAL TRIAL: NCT03290300
Title: A Prospective, Multi-Center, Non-Randomized Study to Evaluate the Quality of Life Impact After Treatment of Nasal Airway Obstruction Using the Aerin Medical Vivaer Stylus
Brief Title: Quality of Life Impact of Nasal Airway Treatment With Aerin Medical Device
Status: Completed | Type: Observational
Sponsor: Aerin Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: TP465
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Results first posted 2019-08-19 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Nasal Obstruction
Keywords: Nasal valve; Nasal airway obstruction; Quality of Life
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long-Term Study Subjects: This cohort will consist of all subjects who were treated with the Vivaer Stylus in the 50-subject TP258 interventional study, who consent to continue to provide quality of life data.
  Interventions: Device: Vivaer Stylus

INTERVENTIONS:
Device: Vivaer Stylus — Previous nasal obstruction treatment with the Aerin Medical Vivaer Stylus
  Other Names: Aerin Medical Device

SUMMARY:
Evaluation of long-term (5-year) quality of life after nasal airway obstruction treatment with the Aerin Vivaer Stylus

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multi-center follow-up study to collect long term quality of life (QOL) data on a cohort of patients who participated in the Aerin Medical TP258 study "A Prospective, Multi-Center, Non-Randomized Study to Evaluate Treatment of Nasal Airway Obstruction Using the Aerin Medical Device". The TP258 study followed subjects out to 26 weeks post-procedure. This QOL study will collect data at 12, 18, 24, 36, 48 and 60 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Received nasal obstruction treatment in Aerin Study TP 258

Exclusion Criteria:

* Unwilling to participate in this long-term study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects in this study will all have completed participation in the TP 258 Nasal Obstruction study.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2022-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wolf, MD, Study Director — Aerin Medical; Ofer Jacobowitz, MD, PhD, Principal Investigator — ENT and Allergy Associates, Middletown, NY
Locations (8):
- United States (8):
  - Central California Clinical Research, Fresno, California
  - Colorado ENT and Allergy, Colorado Springs, Colorado
  - ENT and Allergy Associates, LLP, Oradell, New Jersey
  - ENT and Allergy Associates, LLP, Bayside, New York
  - ENT and Allergy Associates, LLP, Middletown, New York
  - ENT and Allergy Associates, LLP, New Hyde Park, New York
  - Piedmont Ear, Nose and Throat Associates, Winston-Salem, North Carolina
  - Ear, Nose and Throat Associates of Texas, McKinney, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Long-Term Study Subjects: This cohort consisted of subjects who were treated with the Vivaer Stylus in the 50-subject TP258 interventional study (NCT02914236), who consented to continue to provide quality of life data.
  Vivaer Stylus: Previous nasal obstruction treatment with the Aerin Medical Vivaer Stylus
Period: Overall Study
Arm/Group | Long-Term Study Subjects
Started | 39
Completed | 36
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Long-Term Study Subjects
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39
Baseline NOSE Score [Mean (Standard Deviation); unit: units on a scale] — The Nasal Obstruction Symptom Evaluation (NOSE) scale is a validated disease-specific health status outcomes instrument, used to assess severity of nasal obstruction symptoms. Score ranges from 0 to 100. Higher scores indicate increases symptoms/symptom severity.
  Each subject's baseline score was recorded at the beginning of the previous study, TP258.
  units on a scale | 80.8 (10.7)
26-week NOSE Score (end of previous study) [Mean (Standard Deviation); unit: units on a scale] — The Nasal Obstruction Symptom Evaluation (NOSE) scale is a validated disease-specific health status outcomes instrument, used to assess severity of nasal obstruction symptoms. Score ranges from 0 to 100. Higher scores indicate increases symptoms/symptom severity.
  The 26-week NOSE Score was the last score recorded for each subject at the end of the previous study, TP258.
  units on a scale | 24.9 (21.3)
Change in NOSE score from baseline to 26 weeks [Mean (Standard Deviation); unit: units on a scale] — The Nasal Obstruction Symptom Evaluation score is used to assess severity of nasal obstruction symptoms. The NOSE scale ranges from 0 to 100. A positive number reported for the change from baseline indicates an improved outcome.
  units on a scale | 55.9 (23.6)
26-week responder [Count of Participants; unit: Participants] — A "responder" for the prior study, TP258, was defined as a subject having at least a 15-point improvement in NOSE score (NOSE score described previously). The 39 subjects enrolled in this extension study were categorized as responders or nonresponders based on the change in NOSE score between baseline and the final 26-week follow-up of the previous study.
  Participants | 36

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline NOSE Score
Description: Mean change in Nasal Obstruction Symptom Evaluation (NOSE) score from baseline. The NOSE scale ranges from 0 to 100, so a maximum change from baseline would be 100 points. A positive number reported for the change from baseline indicates an improved outcome.
Time Frame: Baseline, 12, 18, 24 months post-procedure
Population: The population evaluated at 12 months was 36, rather than the full 39 participants, since 3 subjects had not completed the consent process until after the 12-month post-procedure evaluation window. By the 24-month follow-up, 3 subjects had been lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Long-Term Study Subjects - 12 Month Data: This cohort consisted of subjects who were treated with the Vivaer Stylus in the 50-subject TP258 interventional study, who consented to continue to provide quality of life data and were enrolled in this study within the 12-month post-procedure window.
- Long-Term Study Subjects - 18 Month Data: This cohort consisted of subjects who were treated with the Vivaer Stylus in the 50-subject TP258 interventional study, who consented to continue to provide quality of life data and provided data within the 18-month post-procedure window.
- Long-Term Study Subjects - 24 Month Data: This cohort consisted of subjects who were treated with the Vivaer Stylus in the 50-subject TP258 interventional study, who consented to continue to provide quality of life data and provided data within the 24-month post-procedure window.
Arm/Group | Long-Term Study Subjects - 12 Month Data | Long-Term Study Subjects - 18 Month Data | Long-Term Study Subjects - 24 Month Data
Number analyzed (Participants) | 36 | 39 | 36
units on a scale | 53.3 (25.2) | 48.1 (30.2) | 53.5 (24.6)
Statistical Analysis 1: Comparison: Long-Term Study Subjects - 12 Month Data vs Long-Term Study Subjects - 18 Month Data vs Long-Term Study Subjects - 24 Month Data; Test type: Other; p < 0.0001, ANOVA — The pre-specified threshold for statistical significance was p<0.05; Repeated measures ANOVA with multiple comparisons to baseline

2. Primary Outcome: Change From Baseline NOSE Score - Long Term Extended Follow-up
Description: as for outcome 1
Time Frame: Update to include Extended Follow up to 36-, 48- months post-procedure
Population: Of the 49 patients in the initial study,39 agreed to participate in follow-up through 24 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 36 Month; Long-Term Study Subjects - 48 Month Data: This cohort consisted of subjects who were treated with the Vivaer Stylus in the 50-subject TP258 interventional study, who consented to continue to provide quality of life data and provided data within the 48-month post-procedure window.
Arm/Group | 36 Month | Long-Term Study Subjects - 48 Month Data
Number analyzed (Participants) | 28 | 28
score on a scale | 32.3 (21.4) | 25.7 (19.1)

3. Primary Outcome: Number and Percentage of Participants With Positive Response on Quality of Life Assessment Items
Description: This 21-item QOL scale was developed by Aerin Medical for this study to assess durability of symptom relief after treatment for nasal obstruction. Each item had 5 possible answers to convey the following responses: very positive, positive, neutral, negative and very negative. For questions 1-14, those who answered "agree or agree strongly" when prompted with "Compared to before I had the Aerin Medical Nasal Procedure, I have experienced..." were considered to have a positive response. For questions 15-18, those who answered "rarely/very rarely/never" when prompted with "Compared to before you had the procedure, how often did you suffer from the following conditions?..." were considered to have a positive response. For questions 19-21, those who answered "less or much less frequently" when prompted with "Compared to the time prior procedure, how often have you used the following to help you with nasal congestion/difficulty breathing?..." were considered to have a positive response.
Time Frame: 12, 18, 24 months post-procedure
Population: Data missing for some questions not answered by subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Long-Term Study Subjects - 12 Month: This cohort consisted of subjects who were treated with the Vivaer Stylus in the 50-subject TP258 interventional study, who consented to provide quality of life data and completed questionnaires 12 months post-procedure
- Long-Term Study Subjects - 18 Month Data: This cohort consisted of subjects who were treated with the Vivaer Stylus in the 50-subject TP258 interventional study, who consented to provide quality of life data and completed questionnaires 18 months post-procedure
- Long-Term Study Subjects - 24 Month Data: This cohort consisted of subjects who were treated with the Vivaer Stylus in the 50-subject TP258 interventional study, who consented to provide quality of life data and completed questionnaires 24 months post-procedure
Arm/Group | Long-Term Study Subjects - 12 Month | Long-Term Study Subjects - 18 Month Data | Long-Term Study Subjects - 24 Month Data
Number analyzed (Participants) | 36 | 39 | 36
Participants
  Q1: Less difficulty falling asleep | 25 | 22 | 28
  Q2: Less waking up at night | 20 | 25 | 25
  Q3: Better sleep throughout the night | 23 | 27 | 26
  Q4: Waking up feeling rested | 18 | 21 | 22
  Q5: Less fatigue during the day: number analyzed (Participants) | 35 | 39 | 36
  Q5: Less fatigue during the day | 20 | 24 | 19
  Q6: Increased productivity | 13 | 16 | 21
  Q7: Increased energy | 18 | 16 | 22
  Q8: Increased ability to focus: number analyzed (Participants) | 36 | 38 | 36
  Q8: Increased ability to focus | 11 | 18 | 22
  Q9: Increased sense of overall well-being | 18 | 21 | 23
  Q10: Less feelings of frustration | 17 | 21 | 18
  Q11: Less feelings of sadness | 12 | 13 | 17
  Q12: Less feelings of embarrassment | 20 | 13 | 16
  Q13:Missing fewer activites with family/friends | 12 | 13 | 17
  Q14: Missing fewer days at work: number analyzed (Participants) | 35 | 37 | 36
  Q14: Missing fewer days at work | 9 | 8 | 15
  Q15: Headaches | 22 | 27 | 28
  Q16: Sinus infections | 28 | 32 | 33
  Q17: Sore throat | 30 | 33 | 30
  Q18: Post nasal drip | 19 | 19 | 21
  Q19: Oral medications | 23 | 19 | 24
  Q20: Nasal sprays | 26 | 20 | 23
  Q21: Nasal breathing strips: number analyzed (Participants) | 34 | 39 | 36
  Q21: Nasal breathing strips | 22 | 27 | 29

ADVERSE EVENTS:
Time Frame: Between 1 and 2 years post-procedure
Description: Physician's office communicated with the subject either in person or by phone at each follow-up point.
Groups:
- Long-Term Study Subjects: This cohort consisted of subjects who were treated with the Vivaer Stylus in the 50-subject TP258 interventional study, who consented to continue to provide quality of life data.
  Vivaer Stylus: Previous nasal obstruction treatment with the Aerin Medical Vivaer Stylus
Arm/Group | Long-Term Study Subjects
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

LIMITATIONS AND CAVEATS:
use of a single-arm design without randomized control, no control of medication usage, and significant patient attrition relative to the primary study. Two nonparticipants were known to have undergone subsequent surgery for nasal obstruction and it is possible that the effectiveness declined in the extended follow-up nonparticipants, although participants and non-participants had similar baseline characteristics and both groups experienced robust NOSE score reductions at 6months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication of study results shall be made in conjunction with the results from all clinical study centers participating in the multicenter study. If results of the multi-center study have not been published in full within 18 months after completion of the study, investigator shall be free to publish results. Investigator agrees to submit all proposed publications to the sponsor at least 60 days prior submission; the company has the right to comment.

DOCUMENTS (2):
  • Study Protocol (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT03290300/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT03290300/SAP_001.pdf